CLINICAL TRIAL: NCT00640601
Title: A Multicentre, Open-label, Prospective Long-term Study Evaluating the Clinical Benefit and Effectiveness of SEROQUEL XR® (Quetiapine Fumarate Extended-Release Tablets) in Subjects With Schizophrenia
Brief Title: Study Evaluating the Clinical Benefit of SEROQUEL XR in Subjects With Schizophrenia
Acronym: SPECTRUM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1443L00025
Record Dates: First submitted 2008-03-17; First posted 2008-03-21 (Estimated); Results first posted 2012-06-22 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Schizophrenia
Keywords: Seroquel; schizophrenia; Extended Release
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Quetiapine Fumarate Extended- Release — Open-label seroquel XR tablets: On Day 1 Patients received 300 mg, on Day 2 600 mg, on Day 3 600-800 mg and between Day 4-168 400-800 mg Seroquel XR, according to clinical judgement of investigator. Dose changes were in 200 mg fixed doses. Investigational product (IP) was supplied in open label wallet blister cards and subjects were instructed to take the IP once daily in the evening.
  Other Names: Seroquel XR®

SUMMARY:
A Multicentre, Open-label, Prospective Long-term Study Evaluating the Clinical Benefit and Effectiveness of SEROQUEL XR® (Quetiapine Fumarate Extended-Release Tablets) in Subjects with Schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent before initiation of any study related procedures.
* Male and female subjects aged 18 to 65 years, inclusive.
* Documented clinical diagnosis meeting the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV) criteria for any of the following: Schizophrenia DSM-IV, catatonic 295.20, disorganised 295.10, paranoid 295.30 and undifferentiated 295.90.
* Outpatient status.
* Subjects who in their own and/or in the Principal Investigator's opinion, consider their ongoing antipsychotic treatment inadequate because of insufficient efficacy, poor tolerance, and/or non acceptability of their actual dosage regimen (eg. b.i.d, t.i.d, etc).
* Monotherapy with current antipsychotic for at least 7 days prior to initiating treatment (ie, cannot be on more than one antipsychotic during the 7 day period prior to initiating study medication). Note: Subjects on a b.i.d regimen of seroquel IR for 7 days prior to enrolment are eligible to participate in the study.
* Female subjects of childbearing potential must have a negative serum pregnancy test at enrolment and be willing to use a reliable method of birth control, ie, barrier method, oral contraceptive, implant, dermal contraception, long-term injectable contraceptive, intrauterine device, or tubal ligation during the study.
* Capable to make treatment decisions, including being able to understand and comply with the requirements of the study, and judged as such by the Principal Investigator.
* Be able to read and write either English or French at a grade 7 proficiency level.

Exclusion Criteria:

* First episode, drug naive schizophrenic subjects.
* Meeting the criteria for any other (than schizophrenia) DSM-IV Axis I diagnosis, concomitant organic mental disorder or mental retardation that in the opinion of the Principal Investigator may interfere with study conduct or interpretation.
* Substance/alcohol dependence or abuse at enrolment [except dependence in full remission (>3 months) and except caffeine and nicotine dependence] as defined by DSM-IV criteria. A urine drug screen will be performed. The Principal Investigator will evaluate the results along with medical history to determine if the patient meets DSM-IV criteria for substance abuse or dependence. However, a single urine toxicology screen for cocaine, heroin, methamphetamine or PCP will lead to exclusion.
* Subjects requiring treatment with another antipsychotic agent than investigational product during study.
* Subjects on seroquel IR once daily.
* Known lack of response to clozapine or treatment with clozapine within 4 weeks prior to enrolment.
* Known intolerance to seroquel IR.
* Subjects requiring treatment with disallowed medication following enrolment into the study.
* Subjects requiring treatment for epilepsy.
* Subjects who pose an imminent risk of suicide or danger to themselves or others, as judged by the Principal Investigator.
* Pregnancy or lactation.
* A thyroid-stimulating hormone (TSH) concentration more than 10% above the upper limit of the normal range of the laboratory used for sample analysis whether or not the patient is being treated for hypothyroidism or hyperthyroidism.
* Use of a depot or long-acting injectable antipsychotic drug within 1 dosing interval before Day 1 of treatment or during treatment.
* Use of drugs that induce or inhibit the hepatic metabolising cytochrome P450 3A4 enzymes within 14 days of the screening assessment period (Day -7 to 0). See Table 5.
* History of idiopathic or drug-induced agranulocytosis.
* A QTc interval longer than 450 msec (calculated using the Fridericia correction for heart rate) or ECG considered to show cardiac abnormality at enrolment as determined by a centrally located, experienced cardiologist, and confirmed by the Principal Investigator as clinically significant.
* Evidence of clinically relevant disease (eg, renal, hepatic, autonomic, endocrine, hematologic or ophthalmologic impairment, significant coronary artery disease, congestive heart failure, cerebrovascular disease, viral hepatitis B or C, acquired immunodeficiency syndrome [AIDS] or cancer) or a clinical finding that is unstable or that, in the opinion of the Principal Investigator, would be negatively affected by the investigational product or that would affect the investigational product.
* Laboratory test results outside the reference range considered by the Principal Investigator to be clinically significant and potentially interfere with the study outcome.
* A patient with Diabetes Mellitus (DM) fulfilling one of the following criteria:

  * Unstable DM defined as HbA1c >8.5% at enrolment. Admitted to hospital for treatment of DM or DM related illness in past 12 weeks.
  * Not under care of physician responsible for patient's DM care.
  * Physician responsible for patient's DM care has not indicated that patient's DM is controlled.
  * Physician responsible for patient's DM care has not approved patient's participation in the study.
  * Has not been on the same dose of oral hypoglycemic drug(s) and/or diet for the four (4) weeks prior to randomisation. For thiazolidinediones (glitazones) this period should not be less than 8 weeks.
  * Taking insulin whose daily dose on one occasion in the past 4 weeks has been more than 10% above or below their mean dose in the preceding 4 weeks.

Note: If a diabetic patient meets one of these criteria the patient is to be excluded even if the treating physician believes the patient is stable and can participate in the study.

* An absolute neutrophil count (ANC) of <1.5 x 109/L
* Inability to accommodate the visit schedule.
* History of non-compliance as judged by the Principal Investigator.
* Previous enrolment in the present study.
* Participation in another clinical study or compassionate use programme within 4 weeks of screening (Day -7 to 0).
* Involvement in the planning and conduct of the study (applies to both AstraZeneca staff or staff at the study site).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2008-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Chue, MD, Principal Investigator — University of Alberta; Willie Early, MD, Study Chair — AstraZeneca
Locations (36):
- Australia (5):
  - Research Site, Garran, Australian Capital Territory
  - Research Site, Newcastle, New South Wales
  - Research Site, Brisbane, Queensland
  - Research Site, Meadowbrook, Queensland
  - Research Site, Dandenong, Victoria
- Canada (29):
  - Research Site, Calgary, Alberta
  - Research Site, Claresholm, Alberta
  - Research Site, Red Deer, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Victoria, British Columbia
  - Research Site, Miramichi, New Brunswick
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Sydney, Nova Scotia
  - Research Site, Belleville, Ontario
  - Research Site, Brantford, Ontario
  - Research Site, Chatham, Ontario
  - Research Site, Cornwall, Ontario
  - Research Site, Greater Sudbury, Ontario
  - Research Site, London, Ontario
  - Research Site, Markham, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Oakville, Ontario
  - Research Site, Orléans, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Gatineau, Quebec
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Rouyn-Noranda, Quebec
  - Research Site, Verdun, Quebec
  - Research Site, Prince Albert, Saskatchewan
  - Research Site, Saskatoon, Saskatchewan
- Research Site, Hong Kong, Hong Kong
- Research Site, Seoul, Korea, South Korea

REFERENCES:
- [Derived] Chue P, Malla A, Bouchard RH, Lessard S, Ganesan S, Stip E, Johnson S, Chen E, Ahn YM, Kim YS, Robinson G, Schweikert C, Gendron A, Eriksson H; SPECTRUM XR Study Group. The long-term clinical benefit and effectiveness of switching to once-daily quetiapine extended release in patients with schizophrenia. Curr Med Res Opin. 2013 Mar;29(3):227-39. doi: 10.1185/03007995.2012.762903. Epub 2013 Jan 22. PMID 23281876

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 331 patients were enrolled across 40 centers in Canada, Australia, Hong Kong and Korea. Out of these 331 enrolled patients, 295 started treatment on seroquel XR. One hundred and eighty three patients completed the 24-week trial.
Pre-assignment Details: Patients had to fulfill criteria for schizophrenia according to Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV) and their current antipsychotic treatment had to be considered inadequate because of insufficient efficacy, poor tolerance, and/or non acceptability of dosing regimen.
Groups:
- Seroquel XR: Open-label seroquel XR tablets: On Day 1 Patients received 300 mg, on Day 2 600 mg, on Day 3 600-800 mg and between Day 4-168 400-800 mg Seroquel XR, according to clinical judgement of investigator. Dose changes were in 200 mg fixed doses. Investigational product (IP) was supplied in open label wallet blister cards and subjects were instructed to take the IP once daily in the evening.
Period: Overall Study
Arm/Group | Seroquel XR
Started | 295 (331 patients enrolled and 295 patients started investigational product (IP))
Completed | 183
Not Completed | 112
Not completed — Adverse Event | 43
Not completed — Withdrawal by Subject | 20
Not completed — Protocol Violation | 6
Not completed — Lack of Efficacy | 16
Not completed — Lost to Follow-up | 9
Not completed — Physician Decision | 8
Not completed — treatment naive, combination therapy | 10

BASELINE CHARACTERISTICS:
Arm/Group | Seroquel XR
Number analyzed (Participants) | 295
Age Continuous [Mean (Standard Deviation); unit: Years] | 37.8 (12.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113
  Male | 182

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Improved Clinical Benefit From Assessment of Clinical Global Impression-Clinical Benefit (CGI-CB) Scale From Baseline to Week 24 or End of Study
Description: Proportional change in CGI-CB score The CGI-CB scale is used to evaluate investigator's global weighted impression of efficacy and interference of adverse events (AEs) from enrolment to every visit. The score ranges from 1 to 10. The lower the score the better the outcome, e.g.: a score of 1 means that there is marked therapeutic effect with no burden of AEs. A score of 10 signifies that the burden of AEs outweighs the therapeutic effect, or no therapeutic effect with high burden of AEs. A change score for each subject will be calculated by subtracting the baseline score from the visit score.
Time Frame: Baseline to 24 weeks (or end of study)
Population: The intention to treat (ITT) population (i.e., all subjects who received at least one dose of the study medication) comprised the population for the analysis (n=295)
Measure: Mean (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Seroquel XR
Number analyzed (Participants) | 295
Percentage of Participants | 56.88 (0.508) [50.8 to 62.8]

2. Secondary Outcome: Change in Clinical Global Impression-Clinical Benefit (CGI-CB) Score
Description: Numerical change in CGI-CB score. The CGI-CB scale is used to evaluate investigator's global weighted impression of efficacy and interference of adverse events (AEs) from enrolment to every visit. The score ranges from 1 to 10. The lower the score the better the outcome, e.g.: a score of 1 means that there is marked therapeutic effect with no burden of AEs. A score of 10 signifies that the burden of AEs outweighs the therapeutic effect, or no therapeutic effect with high burden of AEs. A change score for each subject will be calculated by subtracting the baseline score from the visit score.
Time Frame: Baseline to 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Seroquel XR
Number analyzed (Participants) | 295
units on a scale | 1.41 (3.843)

3. Secondary Outcome: Change in Positive and Negative Syndrome Scale for Schizophrenia (PANSS) Total Score
Description: Change in PANSS total score which includes Positive, Negative and General psychopathology. The PANSS is a 30-item scale where each symptom is rated on a severity scale ranging from 1-7, where 1=absent, 7=extreme). Maximum total score: 210, minimum total score is 30. Seven items are referring to positive symptoms (P1-7), seven items to negative symptoms (N1-7) and 16 items to general psychopathology (G1-16). The assessment prior to start of treatment is considered the baseline assessment.
Time Frame: Baseline to 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Seroquel XR
Number analyzed (Participants) | 295
units on a scale | 10.95 (20.899)

4. Secondary Outcome: Change in Positive and Negative Syndrome Scale for Schizophrenia (PANSS) Positive Scale Score
Description: Change in positive subscale of PANSS. This subscale calculates the sum of the scores in PANSS items P1-P7. (1=absent symptoms, 7=extreme symptoms). Maximum total score: 49, minimum total score: 7.
Time Frame: Baseline to 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Seroquel XR
Number analyzed (Participants) | 295
units on a scale | 2.36 (6.061)

5. Secondary Outcome: Change in Positive and Negative Syndrome Scale for Schizophrenia (PANSS) Negative Scale Score
Description: Change in negative subscale of PANSS. This subscale calculates the sum of the scores in PANSS items N1-N7. (1=absent symptoms, 7=extreme symptoms). Maximum total score: 49, minimum total score: 7.
Time Frame: Baseline to 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Seroquel XR
Number analyzed (Participants) | 295
units on a scale | 3.67 (6.135)

6. Secondary Outcome: Change in Global Assessment Scale (GAS)
Description: Change in GAS score. The GAS is a 100-point single item scale that rates patient's functioning on a hypothetical continuum of mental health to mental illness. The scale values range from 1 to 100 (1=most impaired, 100=healthiest).
Time Frame: Baseline to 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Seroquel XR
Number analyzed (Participants) | 295
units on a scale | 5.54 (14.866)

7. Secondary Outcome: Change in Clinical Global Impression-Severity (CGI-S) Scale
Description: The CGI-S assesses severity of illness which is scored to rate the patient's current clinical state at start of treatment. The scores range from 1 to 7, where 1= normal, not at all ill, while a score of 7=among the most extremely ill of subjects. The change from start of treatment in the severity of illness is calculated by subtracting the score at start of treatment from the visit score. Alleviation of symptom severity will be indicated by a negative change score.
Time Frame: Baseline to 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Seroquel XR
Number analyzed (Participants) | 295
units on a scale | 0.51 (1.174)

8. Secondary Outcome: Change in Clinical Global Impression-Improvement (CGI-I) Scale
Description: Change in CGI-I scale. This scale is the second part of the CGI scale that is scored at Visit 3 to week 24 to observe the patient's change from start of treatment. The scores for the CGI-I subset ranges from 1 to 7 (1=very much improved, 7=very much worse and a score of 4 indicates no change.)
Time Frame: Day 7 - week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Seroquel XR
Number analyzed (Participants) | 295
units on a scale | 0.55 (1.556)

9. Secondary Outcome: Change in Social and Occupational Functioning Assessment Scale (SOFAS)
Description: Change in SOFAS score. The SOFAS is a 100 point single item scale that rates functioning of a patient. The scale values range from 1=most impaired to 100=healthiest individual. The scale also includes a rating point of 0=missing information.
Time Frame: Baseline to 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Seroquel XR
Number analyzed (Participants) | 295
units on a scale | 6.45 (13.820)

10. Secondary Outcome: Change in Safety Measure: Simpson-Angus Scale (SAS)
Description: The Percentage of patients with change in Simpson-Angus Scale (SAS)was calculated. This is a 10 item scale that is rated on a five-point scale where 0=normal and 4=severe symptoms of Extrapyramidal symptoms (EPS) with a focus on parkinsonian symptoms of EPS.
Time Frame: Baseline to 24 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of subjects
Arm/Group | Seroquel XR
Number analyzed (Participants) | 295
Percentage of subjects
  Improved | 46.1
  Unchanged | 43.5
  Worsened | 10.4

11. Secondary Outcome: Change in Barnes Akathisia Rating Scale (BARS)
Description: The Percentage of patients with change in BARS score was calculated. The BARS is a 4 item scale that is rating Extrapyramidal symptoms (EPS) on a 4-point scale for the first three questions and on a 6-point scale for the last question. 0=normal and a higher value represents more pronounced symptoms of EPS. BARS has a focus on the akathisia symptoms of EPS.
Time Frame: Baseline to 24 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Seroquel XR
Number analyzed (Participants) | 295
percentage of subjects
  Improved | 28.1
  Unchanged | 63.7
  Worsened | 8.2

ADVERSE EVENTS:
Arm/Group | Seroquel XR
Serious Adverse Events (participants affected / at risk) | 33/295
Other Adverse Events (participants affected / at risk) | 224
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Seroquel XR (N=295)
Gastritis (Gastrointestinal disorders) | 1
Appendicitis (Infections and infestations) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Acute psychosis (Psychiatric disorders) | 2
Aggression (Psychiatric disorders) | 1
Delusion (Psychiatric disorders) | 2
Delusional Perception (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
Hallucination; Auditory (Psychiatric disorders) | 1
Homicidal Ideation (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Major Depression (Psychiatric disorders) | 1
Psychotic Disorder (Psychiatric disorders) | 8
Schizoaffective Disorder Bipolar Type (Psychiatric disorders) | 1
Schizophrenia (Psychiatric disorders) | 8
Schizophrenia; Disorganised Type (Psychiatric disorders) | 1
Suicidal Behaviour (Psychiatric disorders) | 1
Suicidal Ideation (Psychiatric disorders) | 3
Suicide Attempt (Psychiatric disorders) | 3
Orthostatic Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Seroquel XR
Somnolence (Nervous system disorders) | 53/295
Dizziness (Nervous system disorders) | 43/295
Sedation (Nervous system disorders) | 42/295
Dry Mouth (Gastrointestinal disorders) | 38/295
Anxiety (Psychiatric disorders) | 27/295
Constipation (Gastrointestinal disorders) | 27/295
Headache (Nervous system disorders) | 26/295
Insomnia (Psychiatric disorders) | 24/295
Fatigue (General disorders) | 22/295
Weight Increased (Investigations) | 22/295
Nausea (Gastrointestinal disorders) | 17/295

LIMITATIONS AND CAVEATS:
The open-label design and lack of a placebo group constitute potential limitations. In addition, the small sample size of some of the subgroups may limit conclusions drawn from subgroup analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AstraZeneca shall have a period of 30 days from receipt of the proposed final manuscript for any publication or other disclosure to review it and may within such time require that submission for publication or disclosure of the manuscript be delayed for an additional period of ninety (90) days in order for AstraZeneca to file patent applications.